CLINICAL TRIAL: NCT04750408
Title: Clinical Effects of Nasal High-flow Compared to Oxygen in Acute Viral Illness
Brief Title: NHF vs. COT in Hypoxemic Pandemic Viral Illness
Acronym: HIVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jens Bräunlich (Other)
Responsible Party: Sponsor-Investigator, Jens Bräunlich, Chair Pneumology and Respiratory Medicine, Klinikum Emden
Organization: Klinikum Emden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2021-01-21; First posted 2021-02-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Acute Viral Bronchitis; Hypoxemic Respiratory Failure; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen use (Active Comparator): Patients will use standard oxygen via face mask of nasal prongs as usual care.
  Interventions: Device: Standard oxygen
- NHF use (Experimental): Patients will use NHF instead of oxygen. Oxygen will be supplemented via the NHF flow.
  Interventions: Device: Nasal high-flow

INTERVENTIONS:
Device: Standard oxygen — COT describes the application of low-flow oxygen in any way (Hudson mask, nasal prongs,...).
  Other Names: COT
  Arms: Oxygen use
Device: Nasal high-flow — F is combination of room air supplemented with oxygen can be better patients. This gas mixture will be provided to the patient with a specialized nasal prong.
  Other Names: NHF
  Arms: NHF use

SUMMARY:
The study compares oxygen and NHF in patients with acute viral illness. The duration will be 72h. After them physiological parameters and the outcome will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* acute hyperemic viral illness
* acute hyperemic or hypercapnia respiratory failure

Exclusion Criteria:

* intubation criteria
* indication for NIV therapy
* influences of primary endpoint (rip fracture, lung embolism)
* tracheostomy
* other interventional trials
* noncompliance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
Rox index | 72 hours
  (SpO2/FiO2)/RR = index without a unit, mean Rox-index in the two groups, comparison between the groups (significant differences), physiological parameter, to assess differences between the two groups

SECONDARY OUTCOMES:
paCO2 in mmHg | 72 hours
  physiological parameter, to assess differences between the two groups
pH | 72 hours
  physiological parameter, to assess differences between the two groups
escalation of therapy | 72 hours
  use of noninvasive ventilation, intubation, to assess differences between the two groups
paO2 in mmHg | 72 hours
  physiological parameter, to assess differences between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Jens Bräunlich, MD, Study Chair — chair
Locations (1):
- Klinikum Emden, Emden, Germany

IPD SHARING:
Plan to Share IPD: Yes
original/ raw data
Supporting Information: Study Protocol, ICF
Time Frame: after the end of the study
Access Criteria: on request